Enhancing School-Based Violence Prevention NCT04087772 January 24, 2024



Enhancing School-Based Violence Prevention Regional Superintendent ADDRESS PHONE



Parent Information Letter

January 24, 2024

Dear Parent/Guardian,

We continue to be excited about our partnership with the University of Florida (UF), Medical University of South Carolina (MUSC), and University of South Carolina (USC) on a study funded by the National Institutes of Health to investigate how student health can be improved.

All students who are in 9<sup>th</sup> grade whose middle school was in the study are again being asked to participate in an assessment of the project's impact by filling out surveys that will ask about your child's behavior, and how he or she manages emotions If you would like to view a copy of the questions that your child would be asked, you may do so by contacting (XXX) via the information listed at the top of this form. Students completed this survey in Fall 2021, Spring 2022, and Spring 2023 and we want to ask your child to complete them again in Spring 2024. The survey will take no more than 45 minutes to complete each time. Your child will get to choose if he/she wants to take part on the day that the surveys are given. At the same time, other information will be collected about your child through teacher surveys.

Participation in this study is considered "low risk," however if your child feels uncomfortable about sharing feelings and behaviors on the surveys, he/she may skip any question that they don't want to answer. While we are confident that the study will help us to learn ways to help students feel better and succeed at school, and that what we learn will improve health and learning outcomes in your school district, your child may not benefit directly from participation. The researchers may benefit professionally if the results of the study are presented at meetings or in scientific journals.

All information will be coded with a number so no names are present in any of the documents. Researchers will never see student names and school staff will never see student responses. This means your child's responses and his/her teacher's responses will not be identifiable by school staff or researchers. All de-identified responses will be kept private and stored in locked filing cabinets or in computers with security passwords. At the end of the study, school staff will destroy the list linking student names and survey code numbers; then participant responses will be wholly anonymous.

Your child does not have to take part in the surveys or may stop responding to the surveys at any time. If your child stops completing the survey, there will be no cost or loss of services, or negative outcomes, and the information that he/she already gave us will stay private. If the results of this research are published or presented at scientific meetings, your child's identity will not be disclosed. Researchers will take appropriate steps to protect any information they collect about your child.

If you wish to discuss the information above, please contact (XXX) via the information at the top of this form. If you have any questions regarding your rights as a research subject, please contact the Institutional Review Board (IRBO2) office (XXX) or (XXX) XXX-XXXX).

Do you voluntarily consent to have your child complete these surveys? If so, we will proceed.

If you DO NOT want your child to fill out the surveys, please contact the Project RISE program specialist at your district by calling (XXX) XXX-XXXX or emailing (XXXXXXXX) within two weeks of receiving this letter. If your child did not participate in the Fall 2021 survey at your request they will not be asked to participate again unless you contact the study specialist to enroll them.

Thank you very much for considering participation in PROJECT RISE!

Sincerely,

**SIGNATURE**